CLINICAL TRIAL: NCT00434174
Title: A Phase I Study Investigating the Combination of Everolimus With Pemetrexed in Patients With Advanced Non Small Cell Lung Cancer (NSCLC) Previously Treated With Chemotherapy
Brief Title: Safety of Everolimus and Pemetrexed in Lung Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2112; 2006-002759-34
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2012-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung cancer; Non small cell lung cancer; NSCLC; RAD001; Everolimus; Afinitor; Pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Everolimus; Pemetrexed

ARMS (2):
- everolimus + Pemetrexed - daily (Experimental): Daily treatment
  Interventions: Drug: Everolimus; Drug: Pemetrexed
- everolimus + Pemetrexed - weekly (Experimental): Weekly treatment
  Interventions: Drug: Everolimus; Drug: Pemetrexed

INTERVENTIONS:
Drug: Everolimus — RAD001 will be supplied by Novartis as tablets in 3 different dosage strengths, 2.5, 5 and 10 mg. All proposed dose levels in this study can be given as a combination of these dose strengths.
  Daily doses of 2.5, 5, 7.5 and 10 mg of RAD001 will be given alongside the standard 21-day cycle of pemetrexed.
  Other Names: RAD001; Affinitor
Drug: Pemetrexed — Pemetrexed was supplied to the sites in 500 mg/m2 was administered on Day 1 of each cycle as a 10-minute continuous i.v. infusion in 100mL normal saline

SUMMARY:
This study will evaluate the safety of everolimus in combination with pemetrexed when used as treatment in patients with non small cell lung cancer.

ELIGIBILITY:
Inclusion criteria:

* Lung cancer
* Only one prior regimen of chemotherapy for the treatment of non small cell lung cancer
* Adequate bone marrow function
* Adequate liver function
* Adequate renal function
* Negative serum pregnancy test

Exclusion criteria:

* History of another primary malignancy in the last 5 years
* Having recently received an investigational drug
* Having recently received major surgery of wide field radiotherapy
* Chronic treatment with immunosuppressive therapy, steroids or liver enzyme modulators
* Severe or uncontrolled medical conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Establish feasible dose levels/regimens of everolimus combined with pemetrexed chemotherapy through estimation of the End-of-Cycle 1 DLT rate. | Over 18 weeks of combination treatment

SECONDARY OUTCOMES:
Assess the ability to deliver the standard pemetrexed treatment (relative dose intensity) Assess the pharmacokinetics of everolimus and chemotherapy Evaluate the effect of therapy (RECIST) | Over 18 weeks of combination treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Chair — Novartis
Locations (5):
- Australia (2):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Leuven, Belgium
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Hamburg

REFERENCES:
- See also: Results for CRAD001C2112 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4423